CLINICAL TRIAL: NCT03683459
Title: Safety and Efficacy Study of FemFlow Drug-Eluting Peripheral Balloon Catheter for Lesions With Femoral-popliteal Artery Stenosis or Occlusion: a Prospective, Multi-centre, Objective Performance Criteria Clinical Trial.
Brief Title: Safety and Efficacy Study of FemFlow Drug-Eluting Peripheral Balloon Catheter
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lifetech Scientific (Shenzhen) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEB-01
Record Dates: First submitted 2018-09-20; First posted 2018-09-25 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Femoral Artery Stenosis; Femoral Artery Occlusion; Popliteal Arterial Stenosis; Popliteal Artery Occlusion
Keywords: FemFlow; Drug-eluting peripheral balloon catheter

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- interventional arm (Experimental): Participants will be treated with FemFlow Drug-Eluting Peripheral Balloon Catheter.
  Interventions: Device: FemFlow Drug-Eluting Peripheral Balloon Catheter

INTERVENTIONS:
Device: FemFlow Drug-Eluting Peripheral Balloon Catheter — Medical devices will be applied to the enrolled subjects. The arterial pathway was established, followed by lower limb arteriography, and the auxiliary equipment was selected according to the stenosis of the subject's target lesions, followed by pre-dilation. Patients with residual stenosis ≤70% after pre-dilation and suitable for simple balloon dilation catheter treatment can be enrolled. Select the appropriate size of the experimental drug balloon for expansion, then radiography was used to observe the expansion effect, if necessary, multiple expansion can be conducted, and finally withdraw the instrument and suture the puncture point.

SUMMARY:
A prospective, multi-centre, objective performance criteria clinical trial to evaluate the safety and efficacy of FemFlow Drug-Eluting Peripheral Balloon Catheter manufactured by Lifetech Scientific (Shenzhen) Co., LTD. for lesions with femoropopliteal artery stenosis or occlusion.

DETAILED DESCRIPTION:
This study is a prospective, multi-centre, single-group target value clinical study. Taking the patency rate at 12 months after operation as the primary evaluation index and taking target vascular cavity loss rate at 6 months postoperatively, Rutherford Classification at 12 months postoperatively, the ankle/brachial index (ABI), revascularization rate of target lesions, revascularization rate of target vessels, operating success rate and success rate of surgery as the secondary evaluation indexes to evaluate the efficacy of FemFlow Drug-Eluting Peripheral Balloon Catheter manufactured by Lifetech Scientific (Shenzhen) Co., LTD. for lesions with femoropopliteal artery stenosis or occlusion. Taking the incidence of major adverse events (MAE), adverse events (AE) and instrument defects occurred through the entire trail as the evaluation indexes to evaluate the safety of FemFlow Drug-Eluting Peripheral Balloon Catheter manufactured by Lifetech Scientific (Shenzhen) Company for lesions with femoropopliteal artery stenosis or occlusion. According to statistical hypothesis and sample size calculation, the sample size of this clinical trial was 208 cases. All subjects were followed up 1 month, 6 months and 12 months after treatment with a FemFlow Drug-Eluting Peripheral Balloon Catheter, and data on efficacy and safety were collected. All relevant clinical data are managed and analyzed by the professional data management centre and the statistical centre. End-point events of clinical trials are determined by a specially established third party.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients aged greater than 18 years old and less than 85 years old, regardless of gender；

  2. Patients with peripheral femoral or popliteal artery stenosis (greater than or equal to 70%) or occlusive disease;

  3. Rutherford classification graded 2-5；

  4. The subject or its legal representative can understand the purpose of the study, show sufficient compliance with the test protocol, and sign the informed consent.

Exclusion Criteria:

* 1. Patient with arteritis;

  2. Any acute thrombosis of target vessels requires thrombolysis or thrombectomy, or accepted local or systemic thrombolysis within 48 hours；

  3. Any cerebrovascular accidents within 3 months；

  4. Any unstable coronary heart disease or myocardial infarction within 3 months；

  5. Any important organ failure；

  6. Any known hypersensitivity to heparin, aspirin, clopidogrel, paclitaxel, paclitaxel compounds and contrast agents;

  7. Cannot accept antiplatelet and/or anticoagulation therapy；

  8. Patients with hemorrhagic physical diseases；

  9. Alanine transaminase (ALT) or Aspartate transaminase (AST) were five times higher than the normal upper limit；

  10. Serum creatinine > 2mg/dl (177umol/L)；

  11. Pregnant or lactating woman；

  12. In the absence of intervention, the three lumens of tibialis anterior, tibialis posterior and peroneal artery stenosis or occlusion degree were all >50%；

  13. iliac artery stenosis >50%, or lumen stenosis >50% after treatment (Limited to non-drug-eluting balloon or stent treatment only)；

  14. The guide wire cannot pass through target lesions (Passing through target lesions refers to the head of the guidewire arrive beyond the lesion in the absence of interlayer or perforation)；

  15. Severe calcification at target lesions and should not be treated with balloon dilatation therapy;

  16. Pre-dilation or anticipated severe vascular dissections after dilation;

  17. Residual stricture of >50% or severe current-limiting dissection after pre-dilation is not suitable for simple balloon dilatation catheter treatment;

  18. The total length of target lesions is >200mm, or the reference diameter of the target vessel was >7mm or <3mm;

  19. Life expectancy is less than one year;

  20. Participated in clinical trials of other drugs or instruments at the same time;

  21. Other conditions not suitable for inclusion judged by researchers.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2018-07-18 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Patency rate of the first phase | Postoperative 30 ± 7days
  Target vessel patency is defined as all target lesion lumen stenosis of the target vessel ≤50%. Doppler ultrasonography showed that the peak systolic velocity ratio (PSVR) was ≤ 2.4, which could be considered as the target lesion stenosis ≤50%.

SECONDARY OUTCOMES:
Target vascular cavity loss rate. | Postoperative 180 ± 28days
  Target vascular cavity loss rate (LLL) is defined as the value of the minimum diameter reduction in the segment of target lesions after surgery. Evaluation was performed by lower limb artery digital subtraction angiography (DSA) examination.
Rutherford Classification. | Postoperative 30 ± 7days
  Stage 0 - Asymptomatic Stage 1 - Mild claudication Stage 2 - Moderate claudication - The distance that delineates mild, moderate and severe claudication is not specified in the Rutherford classification, but is mentioned in the Fontaine classification as 200 meters.
  Stage 3 - Severe claudication Stage 4 - Rest pain Stage 5 - Ischemic ulceration not exceeding ulcer of the digits of the foot Stage 6 - Severe ischemic ulcers or frank gangrene
Ankle/brachial index (ABI) | Postoperative 30 ± 7days
  The ankle/brachial index (ABI) is defined as the systolic pressure ratio of the tibialis posterior artery or tibialis anterior artery of the affected limb to the ipsilateral brachial artery when the subject is lying flat.
Revascularization rate of target lesions | Postoperative 30 ± 7days
  Target lesion revascularization was defined as finding target lesion embolism or restenosis (stenosis in diameter of >50%) during follow-up, and additional intervention was required according to clinical symptoms.
Revascularization rate of target vessels | Postoperative 30 ± 7days
  Target lesion revascularization was defined as finding target vessels embolism or restenosis (stenosis in diameter of >50%) during follow-up, and additional intervention was required according to clinical symptoms.
Operating success rate | Intraoperative
  Successful operation is defined as in the course of operation, the peripheral balloon catheter can reach the location of the disease and successfully expand, fail to rupture the balloon, and successfully withdraw.
Success rate of surgery | Intraoperative
  The success of surgery is defined as the residual stenosis rate ≤30% during the operation.

CONTACTS AND LOCATIONS:
Overall Officials: Guowei Fu, Principal Investigator — Fudan University
Locations (18):
- China (18):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Zhongshan Hospital Xiamen University, Xiamen, Fujian
  - The First People's Hospital of Foshan, Foshan, Guangdong
  - Zhongshang People's Hospital, Zhongshan, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Hainan General Hospital, Haikou, Hainan
  - The Central Hospital of Wuhan, Wuhan, Hebei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The First Affiliated Hospital of University of South China, Hengyang, Hunan
  - Shandong Provincial Hospital, Jinan, Shandong
  - Yantai YuHuangDing Hospital, Yantai, Shandong
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality
  - Shanghai Ninth People's Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - Affiliated Hospital of Chengdu University of Traditional Chinese Medicine, Chengdu, Sichuan
  - Tianjing Medical University General Hospital, Tianjin, Tianjin Municipality